CLINICAL TRIAL: NCT04233658
Title: Cynara Scolymus Extract for Treatment of Diabetes Mellitus Type 2, a Pilot Clinical Trial Clinical Study Protocol
Brief Title: Cynara Scolymus Extract for Treatment of Diabetes Mellitus Type 2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stefan Fischli (Other)
Responsible Party: Sponsor-Investigator, Stefan Fischli, Deputy Head Division of Endocrinology and Diabetes, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-17
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — artichoke leaf

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cynara Scolymus (Experimental)
  Interventions: Drug: Cynara Scolymus

INTERVENTIONS:
Drug: Placebo — 3x2 capsules / day
  Arms: Placebo
Drug: Cynara Scolymus — 3x2 capsules / day
  Arms: Cynara Scolymus

SUMMARY:
Edible parts of the artichoke plant (Cynara cardunculus, Cynara scolymus) are traditionally known in folk-medicine for lipid lowering and choleretic effects. Furthermore, antidiabetic effects are described. In the past year's research attributed health promoting effects to the main active compounds chlorogenic acid, luteolin and apigenin. Present literature indicates potential antidiabetic effects by different mechanisms like downregulation of gluconeogenesis, increased GLP-1 secretion and modification of insulin signalling. Up to now only few human clinical trials provide insufficient data to conclude the therapeutic potential of cynara scolymus extract in the treatment of type 2 diabetes.

The primary objective is to evaluate the antidiabetic effect and the mechanisms of glucose lowering by a 12-week treatment with a highly-standardized extract of cynara scolymus in subjects with diabetes mellitus type 2 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old.
* Diagnosis of diabetes mellitus type 2 ≥ 90 days prior to screening
* HbA1c-level between 6.5-9%
* Body mass index of ≥ 28 kg/m2
* Stable daily dose (for at least 30 days) of 1-3 oral antidiabetic drug (metformin, sulfonylurea, SGLT-2 inhibitor, thiazolidinedione or DPP-IV-inhibitor)

Exclusion Criteria:

* Subjects with diabetes mellitus type 1 or history of ketoacidosis,
* Uncontrolled diabetes, defined as fasting plasma glucose ≥20mmol/l or recurrent hypoglycemia (defined as capillary glucose values ≤3.5mmol/l)
* Use of insulin or GLP-1-receptor agonists
* Women wanting to become pregnant
* Pregnant or breast-feeding women
* Known hepatic disorder
* Severe renal insufficiency (GFR ≤30ml/min)
* History of inflammatory bowel disease
* History of gastric bypass or gastric sleeve surgery
* Anticoagulation with vitamin K-antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1c-level from baseline to week 12 | 12 weeks